CLINICAL TRIAL: NCT06587464
Title: Exploring Symptom Profile and Treatment Patterns in Korean HAE Patients Using Digital Patient Diary: A Retrospective Descriptive Study (SPEAKUP Study)
Brief Title: A Study to Explore Hereditary Angioedema (HAE) Symptoms and Treatment Patterns in Korean People
Acronym: SPEAKUP
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-667-4004
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Drug Therapy
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HAE Participants (Type I or II): Participants with HAE type I or II who are prescribed icatibant, enrolled in the patient support program (PSP), and registered in the "MyHAE Story" mobile app will be included and their data will be collected retrospectively from the first documented date of app until the date of the last recorded attack, participant withdrawal, loss to follow-up, or the end of the study, whichever occurs first.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
This study intends to gather information on HAE attack symptoms, how often the attacks occur, and the number of times treatment is required to manage the attacks in Korean people over a period of up to 11 months.

The main aims of this study are the following:

* To describe the patterns of HAE attacks, including how often they occur, where they happen in the body, how severe they are, the time between attacks, and any warning signs that appear before an attack.
* To assess how HAE is treated, particularly looking at how on-demand treatments are used during HAE attacks.
* To learn about the people who suffer from HAE attacks (e.g. age, gender, for how long they have been suffering from HAE, and if they use danazol to manage HAE).

In this study, already existing data will be collected and reviewed from a mobile application called "MyHAE Story". The study will only review data collected as part of the clinical routine practice. The study will not impact the standard medical care and treatment of participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are participants in the OnHeart PSP program.
* Participants who have registered in "MyHAE Story" mobile application.

Exclusion Criteria:

- Participants who neither have made input to at least one attack nor have run the app by clicking 'myHAE story' tab within the Kakaotalk chat message at least once after app registration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HAE type I or II participants who are prescribed icatibant, enrolled in the OnHeart PSP, and registered in and actively utilized mobile app application for at least 1 month will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
HAE Attack Rate | Up to 11 months
  The HAE attack rate will be calculated as a per participant per month (PPPM) rate. The PPPM rate will be calculated by dividing the total number of attacks reported per each HAE participant during their observation periods by their duration of observation periods in months.
Percentage of Participants With HAE Attack Based on Location | Up to 11 months
  Number of participants with HAE attack based on anatomical location (face, throat, arm, hand, abdomen, genital, leg, foot) will be evaluated.
Percentage of Participants With HAE Attack Based on Attack Severity | Up to 11 months
  The HAE attack based on severity will be determined using following definitions: mild (temporarily feels somewhat uncomfortable, swelling is alleviated within 48 hours), moderate (slight disruption in daily life), severe (symptoms that make it impossible to carry out daily life).
Average Time Interval Between HAE Attacks in Days | Up to 11 months
Percentage of Participants With Prodromal Symptom | Up to 11 months
  The presence of prodromal symptoms among participants, a response of "No" indicates the absence of any symptoms and a response of "Yes" suggests the presence of one or more symptoms from the following list will be reported: tight and stinging feeling in the skin, anxiety, nausea, sudden emotional changes, non-pruritic rash, severe fatigue, or other symptoms.

SECONDARY OUTCOMES:
Icatibant-treated HAE Attack Rate | Up to 11 months
  The icatibant-treated HAE attack rate will be calculated as a PPPM rate. The PPPM rate will be calculated by dividing the total number of icatibant-treated attacks reported per each HAE participant during their observation periods by their duration of observation periods in months.
Percentage of Icatibant-Treated HAE Attacks Among All HAE Attacks | Up to 11 months
Number of HAE Attacks Categorized Based on the Icatibant Administration in a Single Attack | Up to 11 months
  The number of icatibant administration in a single attack will be reported as either none, once, or twice.
Number of Participants Categorized Based on Demographic Characteristics | At Baseline
  Number of participants will be reported by their demographic characteristics (age, sex, disease duration and baseline danazol use).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/27c786afd674478b??page=1&idFilter=TAK-667-4004